CLINICAL TRIAL: NCT00130273
Title: Managed Problem Solving: An HIV Adherence Trial
Brief Title: Managed Problem Solving to Increase Treatment Adherence in Individuals With HIV
Acronym: MAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Robert Gross, Associate Professor of Medicine and Epidemiology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH067498 (NIH); R01MH067498 (NIH); DAHBR 9A-ASPG
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Problem Solving; Antiretroviral Therapy, Highly Active; Patient Compliance
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Patient Compliance | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Experimental): Participants will receive managed problem solving for 12 months
  Interventions: Behavioral: Managed problem solving
- 2 (Active Comparator): Participants will receive standard of care for 12 months
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Managed problem solving — Participants in the managed problem solving group will have four study visits and will receive three phone calls for the first 3 months of the study, and one phone call every month for the following 9 months. At each study visit, participants will identify barriers to adherence. During the phone calls, participants will be asked about any steps they have taken to improve their adherence. A medication event monitoring system (MEMS) will be used to assess participants' treatment adherence. MEMS uses microelectronic monitors on the caps of medication bottles to record the timing and frequency of bottle openings. Participants whose adherence has decreased or remained the same at the end of 12 months will be evaluated for regimen changes. Blood collection at the beginning and end of the study will be used to measure viral load and CD4 count.
  Arms: 1
Behavioral: Standard care — Participants will receive standard of care for 12 months.
  Arms: 2

SUMMARY:
This study will determine whether a managed problem solving intervention can help patients with HIV better follow their anti-HIV drug regimen and can control HIV better than the standard of care.

DETAILED DESCRIPTION:
HAART is considered to be the most effective treatment for HIV. However, sustained and consistent adherence to HAART is necessary for long-term success. Issues such as memory problems, lack of social support, medication side effects, depression, and substance abuse can significantly reduce patient adherence to HAART. This study will evaluate the effectiveness of a managed problem solving strategy to increase HAART adherence in patients with HIV. Both treatment-naive and treatment-experienced participants will be recruited for this study.

The treatment part of this study will last 12 months. Participants will be randomly assigned to receive the managed problem solving intervention or standard of care for 12 months. Participants in the managed problem solving group will have 4 study visits and will receive 3 phone calls for the first 3 months of the study, and 1 phone call every month for the following 9 months. At each study visit, participants will identify barriers to adherence. During the phone calls, participants will be asked about any steps they have taken to improve their adherence. A medication event monitoring system (MEMS) will be used to assess participants' treatment adherence. MEMS uses microelectronic monitors on the caps of medication bottles to record the timing and frequency of bottle openings. Participants whose adherence has decreased or remained the same at the end of 12 months will be evaluated for regimen changes. Blood collection at the beginning and end of the study will be used to measure viral load and CD4 count. Follow-up phone interviews will be conducted every year for 3 years after the end of treatment.

Study hypothesis: Managed problem solving will result in better adherence to highly active antiretroviral therapy (HAART) and better virologic control and immunological outcomes at the end of 1 year compared with a control group receiving standard or care.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* HIV infected
* Infection likely to be susceptible to a specific treatment regimen
* Have access to a telephone
* Willing and able to comply with all study requirements

Exclusion Criteria for All Participants:

* Live in a care facility that provides medications on schedule

Inclusion Criteria for Treatment-Experienced Participants:

* Restarting HAART after a treatment interruption of at least 3 months OR after virologic failure with a viral load greater than 1,000 copies/ml
* On a treatment regimen for less than 2 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Improved adherence | Measured at Year 4

SECONDARY OUTCOMES:
Decrease in viral load | Measured at Year 4
Increase in CD4 count | Measured at Year 4

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gross, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gross R, Bellamy SL, Chapman J, Han X, O'Duor J, Palmer SC, Houts PS, Coyne JC, Strom BL. Managed problem solving for antiretroviral therapy adherence: a randomized trial. JAMA Intern Med. 2013 Feb 25;173(4):300-6. doi: 10.1001/jamainternmed.2013.2152. PMID 23358784